CLINICAL TRIAL: NCT01895647
Title: Difference of Muscle Power and Myokine Profile After Upper Limb or Lower Limb Electric Muscle Stimulation in Patients With Severe Sepsis and Acute Respiratory Failure
Brief Title: Effect of Different Electric Muscle Stimulation in Patients With Severe Sepsis and Respiratory Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment and high drop-out rate
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kuang-Hua Cheng, MD, visiting staff of pulmonary medicine, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13MMHIS060
Record Dates: First submitted 2013-06-29; First posted 2013-07-10 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Severe Sepsis; Acute Respiratory Failure; Muscle Hypotonia; Inflammation; Weakness
Keywords: electric muscle stimulation; respiratory failure; sepsis; interleukin 6; interleukin 15
MeSH Terms: conditions — Sepsis; Muscle Hypotonia; Inflammation; Asthenia; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biceps stimulation (Experimental): EMS
  Interventions: Device: EMS
- Quadriceps stimulation (Experimental): EMS
  Interventions: Device: EMS
- Control (No Intervention): Control group without electric muscle stimulation

INTERVENTIONS:
Device: EMS — Electric muscle stimulation with programmed warm-up, stimulation and cool-down in 32 minutes
  Other Names: HELEX 573
  Arms: Biceps stimulation; Quadriceps stimulation

SUMMARY:
Rationale : Electric muscle stimulation reduced critical-illness related weakness in patients with severe sepsis and septic shock. But optimal protocol of the stimulation in unknown.

Hypothesis: Focal muscle contraction may improved the muscle power and have systemic anti-inflammatory via cytokine secretion . The difference of electricity used in upper limb or lower limb stimulation may lead to different effect.

Study design: Stratified randomized parallel control study, comparing Biceps, Quadriceps electric muscle stimulation vs. non-stimulation group.

Participant: adult patients with severe sepsis and acute respiratory failure requiring mechanical ventilation.

Intervention: daily stimulation of bilateral Biceps or Quadriceps by programmed electric devices 32 minutes, 5 days/week

Outcome:

1. Primary outcome: Ventilator-dependent days
2. Secondary outcome: change of hand drip muscle power/interleukin-1b/interleukin-6/interleukin-8/TNF-alpha

DETAILED DESCRIPTION:
Background : Severe sepsis and septic shock remain top cause of admission to intensive care unit. Muscle weakness was found in 70-100% patients with severe sepsis and septic shock because of critical-illness induced polyneuropathy and myopathy. Previous study revealed electric muscle stimulation (EMS) could reduce such muscle weakness and mechanical ventilator-dependent days.

Hypothesis: different electricity may be needed for minimal contraction of upper or lower limb because of their muscle size. Induced muscle contraction may lead to myokine secretion and beneficial metabolic and anti-inflammatory effect. Stimulation on Quadriceps may be better than on Biceps.

Participant: adult(older than 20 years-old) patients with severe sepsis.septic shock and acute respiratory failure post mechanical ventilation.

Design: Stratified ( gender and age >50 years-old) Randomized parallel 3 arms study.

Intervention: Daily stimulation of Biceps of Quadriceps after third days in intensive care unit. Programmed electric stimulation device ( HELEX 573 model, strength aggressive. mode, 45-55Hz 32 minutes per day, voltage 30-70mA)

ELIGIBILITY:
Inclusion Criteria:

* severe sepsis or septic shock patients with acute respiratory failure more than 3 days
* adult patients( age>20 years-old)

Exclusion Criteria:

* skin wound/infection near the site of muscle stimulation
* acute myocardial infarction within 7 days
* pregnant women
* uncontrolled epilepsy
* no spontaneous breath because of central or cervical spinal neuropathy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuang H Cheng, Msc, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biceps Stimulation | Quadriceps Stimulation | Control
Started | 8 | 10 | 7
Completed | 8 | 10 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biceps Stimulation | Quadriceps Stimulation | Control | Total
Number analyzed (Participants) | 8 | 10 | 7 | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 78 [73 to 83] | 78 [73 to 83] | 77.5 [72 to 81] | 78 [72 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 5 | 18
  Male | 3 | 2 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 8 | 10 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Ventilator-dependant Days
Description: Patient days on mechanical ventilator ( Our National Health Insurance provide 21 days for acute intensive care at most)
Time Frame: 21 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Biceps Stimulation | Quadriceps Stimulation | Control
Number analyzed (Participants) | 8 | 10 | 7
days | 6 [5.5 to 7] | 7 [5 to 11] | 6 [6 to 15]

2. Secondary Outcome: Muscle Strength Improvement
Description: muscle power measurement by hand grip digital dynamometer every 2 days
Time Frame: 21 days
Population: The measurement cannot be collected because of the patients' drowsiness or incorporation.
Arm/Group | Biceps Stimulation | Quadriceps Stimulation | Control
Number analyzed (Participants) | 0 | 0 | 0

3. Other Pre Specified Outcome: Inflammatory Cytokine Change
Description: Serum interleukin(IL)-1B, IL-6, IL-8, IL-10, IL-15 and tumor necrosis factor(TNF)-alpha will be measured before/after first section of EMS, and after fifth EMS section.
Time Frame: First 1 week.
Population: The data was not completed because undetected IL-15 in first two samples. No data collection was performed for further samples.
Arm/Group | Biceps Stimulation | Quadriceps Stimulation | Control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The first 2 weeks after EMS applied in the ICU.
Arm/Group | Biceps Stimulation | Quadriceps Stimulation | Control
All-Cause Mortality (participants affected / at risk) | 2/8 | 3/10 | 2/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No